CLINICAL TRIAL: NCT03536039
Title: Monoinstitutional Phase II Trial Addressing Tolerability and Activity of RCHOP Chemoimmunotherapy Preceded by BBB Permeabilization by t-NGR Necrosis Factor in Patients With Relapsed/Refractory Primary Central Nervous System Lymphoma
Brief Title: RCHOP Chemoimmunotherapy Preceded BY BBB Permeabilization by t-NGR Necrosis Factor
Acronym: INGRID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andres J. M. Ferreri (Other)
Collaborators: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor-Investigator, Andres J. M. Ferreri, Principal Investigator, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INGRID
Record Dates: First submitted 2017-07-07; First posted 2018-05-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: CNS lymphoma; BBB permeabilization; R-CHOP; TNF
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human; Rituximab; Doxorubicin; Cyclophosphamide; Vincristine; Prednisone; deltacortene

STUDY DESIGN:
Intervention Model Description: Patients will receive NGR-hTNF at dose of 0.8 mcg/sqm 1 hour before standard R-CHOP (cyclophosphamide-doxorubicin-vincristine-prednisone-rituximab) regimen every 3 weeks for six courses (except for course #1 in which only standard R-CHOP regimen will be administered)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGR-hTNF + R-CHOP (Experimental): Treatment includes one course of conventional R-CHOP followed by 5 courses of conventional R-CHOP (rituximab, Cyclophosphamide, vincristine, doxorubicin, prednisone) in conjunction with intravenous delivery of NGR-hTNF. Chemoimmunotherapy courses will be delivered every 3 weeks; day 22 is to be considered as day 1 of the subsequent course
  Interventions: Drug: NGR-hTNF; Other: RITUXIMAB; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: NGR-hTNF — dose of 0.8 mcg/sqm
Other: RITUXIMAB — dose of 375 mg/mq
  Other Names: mabthera
Drug: Doxorubicin — dose of 50 mg/mq
  Other Names: adriamicina
Drug: Cyclophosphamide — dose of 750 mg/mq
  Other Names: endoxan
Drug: Vincristine — dose of 1.4 mg/mq (max 2 mg)
Drug: Prednisone — 75 mg
  Other Names: deltacortene

SUMMARY:
Patients with primary central nervous system lymphoma (PCNSL) are treated with high-dose-methotrexate-based chemotherapy, which requires hospitalization and extensive expertise to manage related toxicity. Treatment with R-CHOP, the most commonly used combination against aggressive lymphomas, could overcome these difficulties, but CNS bioavailability of related drugs is poor due to their limited capability to cross the blood-brain barrier (BBB). Tumor necrosis factor (TNF) induces selective BBB permeabilization and enhances CNS access of anticancer drugs in animal models. The addition of NGR peptide improves biological properties of TNF, resulting in increased drug availability and antitumor synergistic effect, without increased toxicity. Thus, the addition of NGR-hTNF to R-CHOP may result in improved CNS drug availability and activity in patients with relapsed/refractory PCNSL; this hypothesis is being tested in this ongoing phase II trial called "INGRID". This trial will consider HIV-negative patients (age 18-80 ys; ECOG PS ≤3) with relapsed/refractory PCNSL previously treated with high-dose-methotrexate-based chemotherapy± radiotherapy, and with measurable disease.

DETAILED DESCRIPTION:
There are three planned analyses:

1. An exploratory analysis (proof of principle) on the first 10 enrolled patients. In the case the experimental treatment will be safe and some tumor responses will be recorded, the chairman, after due multidisciplinary discussion, could propose to proceed with an open, non-comparative phase II trial, with overall response rate (complete and partial responses) as primary endpoint. The maximum overall response rate considered of low interest will be 30%, and the minimum response rate considered of interest will be 50%; to demonstrate that difference, a total of 28 patients will be needed (one-sided test; trype I error .10; power .9). Importantly, BBB permeabilization will be investigated using different methods. Variations in tumor microvasculature and vessel permeability will be assessed by DCE- and DSC-MRI. Permeability will be assessed in contrast-enhanced lesions, perilesional areas and normal appearing brain; results will expressed as KTRANS values normalized using contralateral normal appearing white matter, and compared by Wilcoxon Signed Rank Test. Concentrations of R-CHOP drugs were assessed on matched CSF and serum/plasma samples.Moreover, BBB permeability will be also assessed by 99mTc-diethylene-triamine-pentacetic acid (99mTc-DTPA) brain scintigraphy.
2. First of the two stages of Simon Minimax design, where 12 patients will be entered (including the 10 patients of the exploratory phase) and, if at least 4 responses will be observed, the study will be continued until a total of 28 patients will be entered.
3. Second stage of Simon Minimax design: final analysis of activity on the whole series (n=28); the experimental treatment will be declared active if at least 12 responses will be observed.

ELIGIBILITY:
Inclusion criteria

* Histological or cytological diagnosis of (D)LBCL
* Disease exclusively localized into the CNS (brain, meninges, cranial nerves, eyes and/or spinal cord) both at first diagnosis and failure
* Progressive or recurrent disease
* Previous treatment with high-dose-methotrexate-based chemotherapy ± WBRT
* Presence of at least one target lesion, bidimensionally measurable
* Age 18 - 80 years
* ECOG performance status 0-3
* Adequate bone marrow (platelets >75.000/mm3, hemoglobin >8 g/dl, ANC >1.000/mm3), renal (serum creatinine <2 times UNL and creatinine clearance ≥40 mL/min), cardiac (VEF ≥50%), and hepatic (SGOT/SGPT <3 times UNL, bilirubin and alkaline phosphatase <2 times UNL) function.
* Given written informed consent prior to any study specific procedures, with the understanding that the patient has the right to withdraw from the study at any time, without any prejudice. Informed consent signed by a patient's guardian is acceptable if the patient is not able to decide inclusion in the study due to cognitive impairment

5.3 Exclusion criteria

* Known HIV disease or other chronic immunodeficiency
* Patients with positive flow cytometry examination of the CSF, but negative results in CSF conventional cytology, and without any other evidence of CNS disease
* Patients with concomitant extra-CNS disease at presentation or relapse
* Symptomatic coronary artery disease, cardiac arrhythmias not well controlled with medication or myocardial infarction within the last 6 months (New York Heart Association Class III or IV heart disease)
* Any other serious medical condition which could impair the ability of the patient to participate in the trial
* Concurrent treatment with other antineoplastic drugs
* Therapy with PPI (Proton Pump Inhibitors, that may interfere with chromogranine levels, see above). For gastroprotective therapy H2-blockers (i.e. ranitidine) are allowed.
* Pregnant and lactating female patients. Sexually active patients of child bearing potential must implement adequate contraceptive measures during study participation.
* Previous or concurrent malignancies at other sites diagnosed or relapsed within the last 3 years of follow-up. Patients with surgically cured in situ carcinomas and basal cell carcinoma of the skin are allowed.
* Presence of any psycological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2019-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
ORR: CR and PR based on IPCG response criteria | up to 18 weeks
  Activity in terms of overall response rate (ORR): Complete Response (CR) and Partial Response (PR) of R-CHOP21 chemo-immunotherapy preceded by BBBP by NGR-hTNF.

SECONDARY OUTCOMES:
Duration of Response (DOR) | 18 months
  DOR will be assessed for all responsive patients; time to documentation of tumor response to failure
Progression-free survival (PFS) | 12 months
  PFS will be assessed for all treated patients; it is defined as the interval between the time of entry onto trial and failure (relapsing or progressive disease), death from any cause or date of the last visit of follow-up
Overall survival (OS) | 12 months
  OS will be assessed for all enrolled patients; it is defined as the time from entry onto trial until death from any cause or date of the last visit of follow-up.
Tolerability: defined by of grade 3-4 AEs according to NCI CTCAE. | 12 months
  Tolerability will be assessed for all enrolled patients; it is defined by of grade 3-4 AEs according to NCI CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Jose Maria Ferreri, MD, Principal Investigator — San raffaele hospital
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreri AJ, Abrey LE, Blay JY, Borisch B, Hochman J, Neuwelt EA, Yahalom J, Zucca E, Cavalli F, Armitage J, Batchelor T. Summary statement on primary central nervous system lymphomas from the Eighth International Conference on Malignant Lymphoma, Lugano, Switzerland, June 12 to 15, 2002. J Clin Oncol. 2003 Jun 15;21(12):2407-14. doi: 10.1200/JCO.2003.01.135. PMID 12805341
- [Background] Connell JJ, Chatain G, Cornelissen B, Vallis KA, Hamilton A, Seymour L, Anthony DC, Sibson NR. Selective permeabilization of the blood-brain barrier at sites of metastasis. J Natl Cancer Inst. 2013 Nov 6;105(21):1634-43. doi: 10.1093/jnci/djt276. Epub 2013 Oct 9. PMID 24108809
- [Background] Curnis F, Sacchi A, Corti A. Improving chemotherapeutic drug penetration in tumors by vascular targeting and barrier alteration. J Clin Invest. 2002 Aug;110(4):475-82. doi: 10.1172/JCI15223. PMID 12189241
- [Background] Corti A, Curnis F, Rossoni G, Marcucci F, Gregorc V. Peptide-mediated targeting of cytokines to tumor vasculature: the NGR-hTNF example. BioDrugs. 2013 Dec;27(6):591-603. doi: 10.1007/s40259-013-0048-z. PMID 23743670
- [Background] Gregorc V, Santoro A, Bennicelli E, Punt CJ, Citterio G, Timmer-Bonte JN, Caligaris Cappio F, Lambiase A, Bordignon C, van Herpen CM. Phase Ib study of NGR-hTNF, a selective vascular targeting agent, administered at low doses in combination with doxorubicin to patients with advanced solid tumours. Br J Cancer. 2009 Jul 21;101(2):219-24. doi: 10.1038/sj.bjc.6605162. Epub 2009 Jun 30. PMID 19568235
- [Background] van Laarhoven HW, Gambarota G, Heerschap A, Lok J, Verhagen I, Corti A, Toma S, Gallo Stampino C, van der Kogel A, Punt CJ. Effects of the tumor vasculature targeting agent NGR-TNF on the tumor microenvironment in murine lymphomas. Invest New Drugs. 2006 Jan;24(1):27-36. doi: 10.1007/s10637-005-4540-2. PMID 16379040
- [Background] Abrey LE, Batchelor TT, Ferreri AJ, Gospodarowicz M, Pulczynski EJ, Zucca E, Smith JR, Korfel A, Soussain C, DeAngelis LM, Neuwelt EA, O'Neill BP, Thiel E, Shenkier T, Graus F, van den Bent M, Seymour JF, Poortmans P, Armitage JO, Cavalli F; International Primary CNS Lymphoma Collaborative Group. Report of an international workshop to standardize baseline evaluation and response criteria for primary CNS lymphoma. J Clin Oncol. 2005 Aug 1;23(22):5034-43. doi: 10.1200/JCO.2005.13.524. Epub 2005 Jun 13. PMID 15955902
- [Background] Reni M, Zaja F, Mason W, Perry J, Mazza E, Spina M, Bordonaro R, Ilariucci F, Faedi M, Corazzelli G, Manno P, Franceschi E, Pace A, Candela M, Abbadessa A, Stelitano C, Latte G, Ferreri AJ. Temozolomide as salvage treatment in primary brain lymphomas. Br J Cancer. 2007 Mar 26;96(6):864-7. doi: 10.1038/sj.bjc.6603660. Epub 2007 Feb 27. PMID 17325700